CLINICAL TRIAL: NCT02963701
Title: Bioequivalence of a Fixed Dose Combination Tablet Containing 400 mg Ibuprofen and 60 mg Pseudoephedrine-HCl Compared to Two Film Coated Fixed Dose Combination Tablets RhinAdvil® (200 mg Ibuprofen and 30 mg Pseudoephedrine-HCl) Administered in at Least 48 Healthy Male and Female Subjects (Open-label, Randomized, Laboratory Blind, Single Dose, Two-way Crossover, Phase I Trial).
Brief Title: Bioequivalence of a Fixed Dose Combination Tablet Containing 400 mg Ibuprofen and 60 mg Pseudoephedrine-HCl Compared to Two Film Coated Fixed Dose Combination Tablets RhinAdvil(R)(200 mg Ibuprofen and 30 mg Pseudoephedrine-HCl) Administered in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 1024.9
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ibuprofen; Acetaminophen

ARMS (2):
- Ibuprofen+Pseudoephedrine-HCl (Experimental): Fixed dose combination
  Interventions: Drug: Ibuprofen; Drug: Pseudoephedrine-HCl
- Ibuprofen+Pseudoephedrine-HCl (RhinAdvil®) (Active Comparator): Fixed Dose Combination
  Interventions: Drug: Ibuprofen; Drug: Pseudoephedrine-HCl

INTERVENTIONS:
Drug: Ibuprofen — Fixed dose combination
Drug: Pseudoephedrine-HCl — Fixed dose combination

SUMMARY:
Primary objective To demonstrate the bioequivalence of a fixed dose combination tablet containing 400 mg Ibuprofen and 60 mg Pseudoephedrine-HCl vs. RhinAdvil® (2 tablets containing 200 mg Ibuprofen and 30 mg Pseudoephedrine-HCl) as a fixed dose combination tablet with respect to the analytes, ibuprofen and pseudoephedrine.

Secondary objective To assess the bioequivalence of a fixed dose combination tablet containing 400 mg Ibuprofen and 60 mg Pseudoephedrine-HCl vs. RhinAdvil® (2 tablets containing 200 mg Ibuprofen and 30 mg Pseudoephedrine-HCl) as a fixed dose combination tablet with respect to R- and S-ibuprofen (enantiomers of ibuprofen).

ELIGIBILITY:
Inclusion criteria:

* Healthy males and females according to the following criteria:
* Based upon a complete medical history, including physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age ≥21 to ≤50 years
* Minimum weight 50kg - both males and females
* Body Mass Index ≥18.5 to ≤29.9 kg/m2
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to admission to the trial
* Male or female patients. Women of childbearing potential1 must be ready and able to use highly effective methods of birth control per International Committee on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly e.g. implants, injectables, combined hormonal contraceptives, intrauterine device, or surgical sterilisation (including hysterectomy). In addition to this, also a barrier method (e.g. male condom) will be required, if the female is not surgically sterilised. A list of contraception methods meeting these criteria is provided in the patient information. Abstaining from sexual activity (if this is the usual lifestyle of the subject) is considered an acceptable method of birth control.

Exclusion criteria:

* Any finding of the medical examination (including Blood Pressure, Pulse Rate and Electrocardiogram) deviating from normal and of clinical relevance at the discretion of the investigator
* Any evidence of a clinically relevant concomitant disease
* Any relevant Gastrointestinal (e.g. ulcera, hernia, bleedings and spasm), hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Any relevant surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or relevant neurological disorders at the discretion of the investigator
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to drug or its excipients) as judged clinically relevant by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least 1 month or less than 10 half-lives of the respective drug prior to first drug administration
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 14 days prior to randomisation
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking on trial days as judged by the investigator
* Alcohol abuse (average consumption of more than 2 units per day for females and more than 3 units per day for males)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration of the trial drug in this study)
* Excessive physical activities within 1 week prior to randomisation or during the trial
* Any laboratory value outside the reference range that is of clinical relevance at the discretion of the investigator
* Inability to comply with dietary regimen of the study centre
* Unwilling to avoid excessive sunlight exposure
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/corrected QT interval (QTc) within 14 days prior to administration or during the trial, and CYP2C8m substrates such as amiodarone, amodiaquine, paclitaxel, rosiglitazone, pioglitazone and repaglinide or CYP2C9 such as warfarin, tolbutamide, phenytoin, losartan, acenocoumarol within 1 month or six half-lives (whichever is greater)
* A marked baseline prolongation of the QTc B interval (e.g., repeated demonstration of a QTc B interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)

Special exclusion criteria:

* Subjects with history of bronchospasm, rhinitis or urticaria associated with Nonsteroidal anti-inflammatory drug (NSAID) - Asthma
* Risk of or manifested narrow-angle glaucoma
* Risk of urinary retention due to urethro-prostatic diseases / prostatic enlargement
* Subjects with the rare hereditary problems of fructose intolerance, glucose-galactose malabsorption or sucrase isomaltase deficiency
* Regular treatment with any systemically available medication (except hormonal contraceptives and hormonal replacement therapy e.g. estrogens, L-thyroxine)
* Subjects, who report a frequent occurrence of migraine attacks
* For female subjects of childbearing potential only:

Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 2 months after study completion

* No adequate contraception during the study including three months before first dosing until 2 month after study completion.
* Lactation

Administrative reasons:

* Subjects suspected or known not to follow instructions
* Subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the study

The exclusion criteria are chosen to assure that subjects with specific risks for administration of the investigational medicinal products and subjects with conditions, which may have an impact on pharmacokinetic parameters, cannot be included

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Bloemfontein Early Phase Clinical Unit, PAREXEL International (South Africa), Bloemfontein, South Africa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was an Open-label, randomised, laboratory blind, single dose, two-way crossover, Phase I trial. A total of 56 healthy male and female subjects were randomised in the trial. Subjects were assigned randomly to one of two treatment sequences (Test-Reference, Reference-Test), before first drug administration.
Groups:
- Treatment Sequence 1 (T-R): Treatment sequence (Test-Reference): The subjects were administered orally under fasting condition first with Test product: Ibuprofen 400 milligram and Pseudoephedrine-HCl 60 milligram fixed dose combination film coated tablet and then with Reference product: 2 x RhinAdvil® (Ibuprofen 200 milligram and Pseudoephedrine-HCl 30 milligram fixed dose combination film coated tablets). Treatments were separated by a washout period of at least 5 days.
- Treatment Sequence 2 (R-T): Treatment sequence (Reference-Test): The subjects were administered orally under fasting condition first with Reference product : 2 x RhinAdvil® (Ibuprofen 200 milligram and Pseudoephedrine-HCl 30 milligram fixed dose combination film coated tablets) and then with Test product: Ibuprofen 400 milligram and Pseudoephedrine-HCl 60 milligram fixed dose combination film coated tablet. Treatments were separated by a washout period of at least 5 days.
Period: Period 1 (Including Washout) (2 Days)
Arm/Group | Treatment Sequence 1 (T-R) | Treatment Sequence 2 (R-T)
Started | 28 | 28
Completed | 27 (One subject withdrawn from the study after period 1) | 28
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2 (2 Days)
Arm/Group | Treatment Sequence 1 (T-R) | Treatment Sequence 2 (R-T)
Started | 27 | 28
Completed | 27 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were calculated on Safety Population. All subjects who received at least one dose of study medication were included in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 (T-R) | Treatment Sequence 2 (R-T) | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.5 (6.77) | 29.2 (8.03) | 28.8 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity data was not collected as per protocol.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 20 | 21 | 41
    White | 7 | 6 | 13
    More than one race | 0 | 0 | 0
    Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to Time of Last Quantifiable Time Point (tz) of Ibuprofen. (AUC0-tz)
Description: This endpoint calculates area under the concentration-time curve of Ibuprofen in plasma over the time interval from 0 to the time of last quantifiable time point.
Time Frame: Samples were collected Pre-dose and at 0:10, 0:20, 0:30, 0:45, 1:00, 1:15, 1:30, 1:45, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 30:00 hours post dose.
Population: Pharmacokinetic Population (PK Set): All treated subjects that provided observations for both periods for at least one primary endpoint evaluable and without any major protocol deviation thought to interfere with the absorption, distribution, metabolism, and excretion of the compound to be measured were included in the PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nano gram per milliliter (h*ng/mL)
Groups:
- Reference Product (R): Subjects were orally administered with RhinAdvil® (Ibuprofen 200 mg and Pseudoephedrine-HCl 30 mg fixed dose combination film coated tablet) (2 tablets)
- Test Product (T): Subjects were orally administered with Ibuprofen 400 mg and Pseudoephedrine-HCl 60 mg fixed dose combination film coated tablet (1 tablet)
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
Hour nano gram per milliliter (h*ng/mL) | 140500 (23.66) | 139300 (19.30)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — A claim of bioequivalence was made if the 90% confidence interval (CI) of the geometric means of T/R ratio was contained in the pre-defined acceptance range of 80.00% to 125.00%; ANOVA; Results are based on ANOVA model on the logarithmic scale including fixed effects for sequence, subject nested within sequence, period and treatment; T/R Ratio (%) = 99.16, 90% CI 2-sided [96.52 to 101.89], Standard Deviation 8.49 — The estimated parameter was the adjusted geometric mean ratios (%) of Test and Reference products. The parameter dispersion type (Standard Deviation) was actually the intra-individual geometric coefficient of variation (%)

2. Primary Outcome: Maximum Concentration of Ibuprofen in Plasma (Cmax).
Description: This outcome is maximum measured concentration of the Ibuprofen in plasma
Time Frame: Samples were collected pre dose and at 0:10, 0:20, 0:30, 0:45, 1:00, 1:15, 1:30, 1:45, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00 and 30:00 hours post dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nano gram per milliliter (ng/mL)
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
Nano gram per milliliter (ng/mL) | 33580 (26.16) | 29940 (20.80)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 89.16, 90% CI 2-sided [83.88 to 94.76], Standard Deviation 19.28 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From 0 to Time of Last Quantifiable Time Point (tz) of Pseudoephedrine (AUC0-tz).
Description: This endpoint calculates area under the concentration-time curve of Pseudoephedrine in plasma over the time interval from 0 to the time of last quantifiable time point.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
h*ng/mL | 2547 (22.22) | 2540 (22.45)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 99.75, 90% CI 2-sided [95.73 to 103.95], Standard Deviation 12.96 — The estimated parameter was the adjusted geometric mean ratios [%] of Test and Reference products. The parameter dispersion type (Standard Deviation) was actually the intra-individual geometric coefficient of variation [%]

4. Primary Outcome: Maximum Concentration of Pseudoephedrine in Plasma (Cmax).
Description: This outcome is maximum measured concentration of the Pseudoephedrine in plasma
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
ng/mL | 320.4 (22.09) | 327.4 (25.28)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 102.16, 90% CI 2-sided [97.30 to 107.27], Standard Deviation 15.37 — The estimated parameter was the adjusted geometric mean ratios [%] of Test and Reference products. The parameter dispersion type [SD] was actually the intra-individual geometric coefficient of variation [%]

5. Secondary Outcome: Area Under the Concentration-time Curve of Ibuprofen in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞).
Description: This endpoint calculates area under the concentration-time curve of Ibuprofen in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
h*ng/mL | 143000 (22.88) | 141600 (18.72)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 98.97, 90% CI 2-sided [96.44 to 101.57], Standard Deviation 8.13 — The estimated parameter was the adjusted geometric mean ratios (%)of Test and Reference products. The parameter dispersion type (Standard Deviation) was actually the intra-individual geometric coefficient of variation (%)

6. Secondary Outcome: Area Under the Concentration-time Curve of Pseudoephedrine in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞).
Description: This endpoint calculates area under the concentration-time curve of Pseudoephedrine in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
h*ng/mL | 2622 (23.07) | 2614 (23.65)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 99.67, 90% CI 2-sided [95.48 to 104.04], Standard Deviation 13.50 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: AUC0-tz of R-Ibuprofen
Description: This endpoint calculates area under the concentration-time curve of R-Ibuprofen in plasma over the time interval from 0 to the time of last quantifiable time point.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
h*ng/mL | 68520 (28.08) | 65760 (21.55)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 95.96, 90% CI 2-sided [91.70 to 100.40], Standard Deviation 14.27 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: AUC0-∞ of R-Ibuprofen
Description: This endpoint calculates area under the concentration-time curve of R-Ibuprofen in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
h*ng/mL | 69420 (27.76) | 66740 (21.51)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 96.12, 90% CI 2-sided [91.92 to 100.51], Standard Deviation 14.06 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Cmax of R-Ibuprofen
Description: This outcome is maximum measured concentration of the R-Ibuprofen in plasma
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
ng/mL | 18630 (29.34) | 16910 (21.98)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 90.83, 90% CI 2-sided [84.87 to 97.21], Standard Deviation 21.49 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: AUC0-tz of S-Ibuprofen
Description: This endpoint calculates area under the concentration-time curve of S-Ibuprofen in plasma over the time interval from 0 to the time of last quantifiable time point.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
h*ng/mL | 70290 (24.90) | 71610 (23.25)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 101.86, 90% CI 2-sided [99.33 to 104.46], Standard Deviation 7.89 — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: AUC0-∞ of S-Ibuprofen
Description: This endpoint calculates area under the concentration-time curve of S-Ibuprofen in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
h*ng/mL | 72270 (23.84) | 73460 (22.21)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 101.65, 90% CI 2-sided [99.40 to 103.95], Standard Deviation 7.01 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Cmax of S-Ibuprofen
Description: This outcome is maximum measured concentration of the S-Ibuprofen in plasma
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
ng/mL | 15050 (22.28) | 13020 (22.36)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; T/R Ratio (%) = 86.53, 90% CI 2-sided [82.03 to 91.28], Standard Deviation 16.85 — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: S/R-ibuprofen Ratio for AUC0-tz
Description: AUC0-tz S-ibuprofen / AUC0-tz R-ibuprofen
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Reference Product (R) | Test Product (T)
Number analyzed (Participants) | 55 | 55
Ratio | 1.026 (23.26) | 1.089 (23.30)
Statistical Analysis 1: Comparison: Reference Product (R) vs Test Product (T); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio (%) = 106.17, 90% CI 2-sided [101.30 to 111.26], Standard Deviation 14.77 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From first drug administration till 7 days after last drug administration; up to 14 days
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have to have a causal relationship with this treatment.
  All subjects who received at least one dose of study medication were included in the safety population.
Arm/Group | Reference Product (R) | Test Product (T)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT02963701/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT02963701/SAP_001.pdf